CLINICAL TRIAL: NCT04826263
Title: Comparison of the Effectiveness of Low-level Laser Therapy and Extracorporeal Shock Wave Therapy in Plantar Fasciitis Treatment
Brief Title: Comparison of the Effectiveness of LLLT and ESWT in Plantar Fasciitis Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Halit SELÇUK, Principal Investigator, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-36
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Plantar Fascitis
Keywords: ESWT; LLLT; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Low-Level Light Therapy; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT Group (Experimental): The patients in the ESWT group will receive ESWT treatment and a home exercise program.
  Interventions: Other: Home Exercise Program; Other: Extracorporeal Shockwave Therapy (ESWT)
- LLLT Group (Experimental): The patients in the LLLT Group will receive LLLT treatment and a home exercise program.
  Interventions: Other: Home Exercise Program; Other: Low-Level Laser Therapy (LLLT)

INTERVENTIONS:
Other: Home Exercise Program — All patients will be instructed to follow a home exercise program for 3 weeks. Patients will be informed about the exercises by giving an exercise sheet describing the exercises and an exercise diary prepared to mark the days they exercise. The home exercise program will include previously recommended exercises such as Achilles tendon and plantar fascia stretching and toe curl exercises. Patients will be instructed to perform these exercises 10 repetitions each and 3 times per day for three weeks.
Other: Low-Level Laser Therapy (LLLT) — Patients in the LLLT group will receive gallium-aluminum-arsenide (Ga-Al-As) low-level laser treatment with Chattanooga Vectra Genisys Transport model (Chattanooga Group) with a wavelength of 850 nm and a power of 100 mW. The LLLT treatment will be applied 3 times a week, a total of 10 sessions. A maximum energy density of 5.6 j/cm2 will be reached by delivering a continuously increasing dose of energy to each tender spot for one minute. The LLLT will be performed with patients in the prone position and will be applied to 5 points on the plantar fascia by positioning the laser head perpendicular to the treatment area.
  Arms: LLLT Group
Other: Extracorporeal Shockwave Therapy (ESWT) — Patients in the ESWT group will receive treatment with a radial ESWT system (EMS Swiss Dolor Clast), which transforms kinetic energy into a shock wave, which is then applied to the target tissue with pressure varying from 1 to 10 bar and penetrating up to 40 mm. The ESWT treatment will be administered to the patients once a week for three weeks, for a total dose of 2000 mJ/mm2 pulse per application. ESWT will be applied to the patients in prone position with their foot inverted. Ultrasound gel will be applied to the patient's heel The area of tenderness will be palpated and 1000 shock wave impulses were applied to this area, and 1000 pulses will be applied over the plantar fascia.
  Arms: ESWT Group

SUMMARY:
The aim of this study is to compare the efficacy of extracorporeal shock wave therapy (ESWT) and low-level laser therapy (LLLT) in terms of pain, disability, activity limitation, gait speed, and cadence in patients with plantar fasciitis (PF).

ELIGIBILITY:
Inclusion Criteria:

* Experience pain on the medial tuberosity or medial process of plantar fascia within the past one month
* Diagnosed with plantar fasciitis

Exclusion Criteria:

* arthritis in the foot or ankle
* Cardiac arrhythmia or pacemaker
* Previous foot or ankle surgery
* Cancer or tumor, acute trauma
* BMI over 40 kg/m2
* Corticosteroid injection in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-04-03 (Estimated); Primary Completion 2021-05-10 (Estimated); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
Foot Function Index (FFI) | It will be reported at baseline
  FFI is a valid and reliable self-administered questionnaire that can evaluate the pain, activity limitation, and disability caused by foot and ankle disorders. A modified version of the Foot Function Questionnaire developed by Venditto et al. will be used for the study, which comprises 17 items (17-IFFI) separated into three subscales; pain (5 items), disability (9 items), and activity limitation (3 items). The VAS in the original version has been substituted with the Numerical Rating Scale (NRS) which is an 11-point scale from 0 to 10. The modified version of FFI has been reported to be a reliable and valid scale and its use has been recommended for musculoskeletal foot and ankle disorders including plantar fasciitis.
Foot Function Index (FFI) | It will be reported at the end of treatment (3 weeks)
  FFI is a valid and reliable self-administered questionnaire that can evaluate the pain, activity limitation, and disability caused by foot and ankle disorders. A modified version of the Foot Function Questionnaire developed by Venditto et al. will be used for the study, which comprises 17 items (17-IFFI) separated into three subscales; pain (5 items), disability (9 items), and activity limitation (3 items). The VAS in the original version has been substituted with the Numerical Rating Scale (NRS) which is an 11-point scale from 0 to 10. The modified version of FFI has been reported to be a reliable and valid scale and its use has been recommended for musculoskeletal foot and ankle disorders including plantar fasciitis.
Gait Speed | It will be reported at baseline (5 minutes after the FFI)
  Patients will be instructed to walk a 25 meters corridor back and forth for 4 times (100 m total). Patients will be instructed to walk as quickly as possible but running will not be allowed. The subjects walking time will be recorded in seconds. Gait speed will be measured by dividing the 100 meters distance by the patients' walking time.
Gait Speed | It will be reported at the end of treatment (3 weeks) (5 minutes after the FFI)
  Patients will be instructed to walk a 25 meters corridor back and forth for 4 times (100 m total). Patients will be instructed to walk as quickly as possible but running will not be allowed. The subjects walking time will be recorded in seconds. Gait speed will be measured by dividing the 100 meters distance by the patients' walking time.
Cadence | It will be reported at baseline (5 minutes after the FFI)
  Patients will be instructed to walk a 25 meters corridor back and forth for 4 times (100 m total). Patients will be instructed to walk as quickly as possible but running will not be allowed. Cadence will be measured by the number of steps in the walking test.
Cadence | It will be reported at the end of treatment (3 weeks) (5 minutes after the FFI)
  Patients will be instructed to walk a 25 meters corridor back and forth for 4 times (100 m total). Patients will be instructed to walk as quickly as possible but running will not be allowed. Cadence will be measured by the number of steps in the walking test.

IPD SHARING:
Plan to Share IPD: No